CLINICAL TRIAL: NCT04460014
Title: Reducing Intrusive Memories After Trauma Via a Simple Cognitive Intervention During COVID-19 in Hospital Staff: "EKUT-P" (Enkel Kognitiv Uppgift Efter Trauma Under COVID-19 - sjukvårdspersonal) - A Randomized Controlled Trial (RCT)
Brief Title: Simple Cognitive Task Intervention After Trauma During COVID-19 In Hospital Staff EKUT-P RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Emily Holmes, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-03085
Record Dates: First submitted 2020-07-06; First posted 2020-07-07 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Intrusive Memories of Traumatic Event(s); Post Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder; Digital Intervention; Intrusive Memories of Traumatic Event(s)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple cognitive task intervention (Experimental): Session 1: A memory cue followed by playing the computer game "Tetris" (e.g. on own smartphone) with mental rotation instructions.
  Options to engage in self-administered/guided booster sessions per intrusive memory.
  Interventions: Behavioral: Simple cognitive task intervention
- Attention placebo (Placebo Comparator): Session 1: Digital activity for same amount of time (e.g. listening to podcast on own smartphone).
  Interventions: Behavioral: Attention Placebo

INTERVENTIONS:
Behavioral: Simple cognitive task intervention — Session 1: A memory cue followed by playing the computer game "Tetris" (e.g. on own smartphone) with mental rotation instructions.
  Options to engage in self-administered/guided booster sessions per intrusive memory.
  Arms: Simple cognitive task intervention
Behavioral: Attention Placebo — Session 1: Digital activity for same amount of time (e.g. listening to podcast on own smartphone).
  Arms: Attention placebo

SUMMARY:
This research study is designed to investigate the effects of a remotely delivered simple cognitive task (a memory cue followed by playing the computer game "Tetris" with mental rotation instructions) on intrusive memories ("flashbacks") and other symptoms after a traumatic event(s). Hospital staff who experienced a work-related traumatic event(s) during the COVID-19 pandemic will be randomly allocated to either the simple cognitive task intervention or control. Randomization to assigned intervention occurs on Day 1, after completion of baseline measures (note: baseline measures are not used in randomization process). Baseline measures include questionnaires on Day 1 and an intrusive memory diary during the previous week (Week 0). Participants will be followed up at one week and one month, and where possible 3 and 6 months. It is predicted that participants given the simple cognitive task intervention will develop fewer intrusive memories, less severe related clinical symptoms, and will show higher functioning (e.g. at work) than those who are not. This will inform the future development of a simple technique to prevent distressing psychological symptoms after a traumatic event(s). Implementation and training aspects regarding remote recruitment and intervention delivery in a hospital context will also be explored. Participants use e.g. their smartphone for part of the intervention in the study.

DETAILED DESCRIPTION:
This is a Randomised Controlled Trial informed by prior feasibility and pilot work (ClinicalTrials.gov IDs: NCT03509792, NCT04185155). The primary outcome is the number of intrusive memories of the traumatic event(s) (week 5). The intervention is delivered remotely (e.g. via smartphone) with potential remote support (e.g. by phone) to medical staff in Swedish hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Clinical work during the COVID-19 pandemic in hospital and care facilities (e.g. ICU, ambulance, intermediate care, ward)
* Experienced at least one traumatic event in relation to their clinical work as health care staff during the COVID-19 pandemic
* This/these event(s) at work meet(s) the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM5) criterion A for Posttraumatic Stress Disorder (PTSD): exposure to actual or threatened death, serious injury, or sexual violence by "Directly experiencing the traumatic event(s)" or "Witnessing, in person, the event(s) as it occurred to others"
* The traumatic event(s) occured since the start of the COVID-19 pandemic
* Report memory of the accident
* Fluent in spoken and written Swedish
* Alert and orientated
* Have sufficient physical mobility to use their smartphone
* Willing and able to provide informed consent and complete study procedures
* Willing and able to be contacted while the study is ongoing
* Have access to an internet enabled smartphone
* Experiences distressing intrusive memories (of a traumatic event in relation to their work as health care staff during the COVID-19 pandemic)
* Has experienced at least two such intrusive memories of a work-related traumatic event during the week before inclusion/exclusion
* Able and willing to briefly write down these intrusive memories (without going into any detail)

Exclusion Criteria:

* Loss of consciousness of > 5 minutes in relation to the traumatic event
* Current intoxication during the traumatic event or in relation to study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories of traumatic event(s) | Week 5
  Number of intrusive memories of traumatic event(s) recorded by participants in a brief diary daily (morning, afternoon, evening and night) for 7 days.

SECONDARY OUTCOMES:
Number of intrusive memories of traumatic event(s) | Week 0 and Week 1
  Number of intrusive memories of traumatic event(s) recorded by participants in a brief diary daily (morning, afternoon, evening and night) for 7 days.
Intrusion questionnaire - frequency item | Baseline (Day 1), Week 1 and 5 and 1, 3, and 6 month follow-up
  A single item measuring the frequency of intrusive/unwanted memories of the traumatic event(s) in the previous week on a 7-point scale (from "never" to "many times a day", with a follow-up question to specify the number if necessary) that will be used as a convergent measure for medical hospital staff who may face time constraints completing the diary.
Intrusion questionnaire - characteristics | Baseline (Day 1), One week and 1, 3, and 6 month follow-up
  5 self-rated items measuring the characteristics of intrusive/unwanted memories in the previous week.
  The level of distress, nowness, reliving, disconnectedness and whether different triggers are associated with the intrusive/unwanted memories of the traumatic event(s) are measured on a 101-point scale (from 0 to 100). Higher scores indicate more intrusive/unwanted memories, higher levels of distress/nowness/reliving/disconnectedness and a greater number of different triggers.
Impact of Event Scale - Revised (IES-R): Degree of subjective distress of post-trauma intrusion and avoidance symptoms | Baseline (Day 1), One week and 1, 3, and 6 month follow-up
  Self-report measure that assesses subjective distress after a traumatic event (with reference to study event[s]) in the last week. Here we include the intrusion subscale (8 items) and the avoidance subscale (8 items). Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Subscale scores are calculated for the Intrusion or Avoidance items summed (ranging from 0 to 32 each). Higher scores indicate worse outcome.
Posttraumatic Stress Disorder Checklist 5 (PCL-5) short version | Baseline (Day 1), One week and 1, 3, and 6 month follow-up
  The PCL-5 short version is an 8-item self-report measure that assesses current symptoms of post-traumatic stress disorder in the last month [Baseline (Day 1), 1, 3, and 6 month follow-up] and in the last week (One week). Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The PCL-5 short version yields a total symptom severity score which ranges from 0 to 32. Subscale symptom severity scores for DSM-5 symptom cluster B - intrusion symptoms (items 1-2), cluster C - avoidance (items 3-4), cluster D - negative alterations in cognitions and mood (items 5-6), and cluster E - alterations in arousal and reactivity (items 7-8). Higher scores indicate worse severity.
Characteristics of intrusive trauma memories | Baseline (Day 1), Week 1 and week 5
  2 self-rated items measuring the level of distress and vividness associated with the intrusions (11 point scales from 0 to 10) rated within the diary at baseline (Day 1), week 1 and week 5. High scores indicate higher level of distress/vividness.

OTHER OUTCOMES:
Self-rated concentration disruption associated with intrusive memories | Baseline (Day 1), Week 1 and Week 5, 1, 3, and 6 months follow-up
  Two items measuring the level of concentration disruption associated with the intrusions (11 point scale from 0 to 10) and the duration of disruption (< 1 min, 1-5 min, 5-10 min, 10-30 min, 30-60 min, > 60 min). High scores indicate higher level of concentration disruption and longer duration of disruption.
Concentration and memory difficulties | 6 month follow-up
  Eleven items assess the extent of concentration and memory difficulties during the previous four weeks, using a 5-point scale (1 'Virtually every day' to 5 'Never'). Total scores range from 11 to 55; higher scores indicate less concentration and memory difficulties.
Self-rated functioning and social support ratings | Baseline (Day 1), One week, 1, 3, and 6 month follow up
  3 bespoke items including a question on impact on work-related functioning, and one on daily functioning in other areas associated with the intrusions and a question on perceived social support after the traumatic event. All items are rated on an 11-point scale (from 0 "none"; 5 "some"; 10 "extreme/much"). Higher scores indicate higher level of functional impairment/perceived social support.
Appraisals of intrusive memories | Baseline (Day 1), One week, 1, 3, and 6 month follow-up
  6 self-report items (11-point scale from 0 to 100) measuring appraisals of intrusions on two subscales: psychological problems (items 1-3) and negative self-evaluations (items 4-6). Items for each subscale will be summed. Possible subscale scores range from 0 - 300, with higher values indicative of worse appraisals.
Self-rated sleep ratings | Baseline (Day 1), one week and 1, 3, and 6 month follow-up
  Two self rated items: Item 1 measures the extent of being troubled by poor sleep (with reference to study event) on a 5 point scale (from not at all to very much), and item 2 measures the number of nights in the week with sleep problems on a 5 point scale (from 0-1 to 5-7 nights). Each 5-point scale is reverse scored (4 - 0) then summed. Possible total scores range from 0 - 8, with higher values indicative of better sleep.
Self Rated Health (SRH) rating | Baseline (Day 1), one week, and 1, 3, and 6 month follow-up
  A single item measuring perceived health status on a seven-point scale (from very good to very bad). The scale is reverse scored. High scores indicate good outcomes.
Questions related to work situation | Baseline (Day 1), One week, 1, 3, and 6 month follow-up
  3 free text response field questions (e.g. which type of health care do you work with right now?) at Day 1 and two free text response field questions on whether the work situation changed and if yes, how, at one week, 1, 3, and 6 month follow-up.
Sick leave | Baseline (Day 1), One week, 1, 3, and 6 month follow-up
  2 bespoke items measuring the total number and the number of full work days on sick leave because of reason for seeking health care. Higher numbers indicate more sick leave.
Stress and Energy Questionnaire (SEQ) - Stress subscale | Baseline (Day 1), One week, 1, 3, and 6 month follow-up
  3 items measuring the frequency of feeling stressed, pressured, tensed at work during the previous week on a 5-point scale (from "never" to "several times per day"). Item scores are summed. Higher scores indicate higher levels of stress. Further, a single item measuring difficulties to let go of work-related thoughts during leisure time (from "very rarely or never" to "very often or always") and a single question about whether the above mentioned difficulties are because of intrusive memories with a yes/no response.
Scale of Work Engagement and Burnout (SWEBO) - Burnout subscale | Baseline (Day 1) and 6 month follow-up
  9 self-report items (4-point scale from 1 "not at all" to 4 "all the time") measuring symptoms of burnout on three subscales: Exhaustion (items 1-3), disengagement (items 4-6) and inattentiveness (items 7-9). Subscale scores will be the mean of all items per subscale, the total burnout score will be the mean of all items (ranging from 1-4) with higher scores indicative of higher levels of exhaustion/disengagement/inattentiveness/burnout.
Moral stress at work | Baseline (Day 1), One week, 1, 3, and 6 month follow-up
  5 self-report items measuring moral stress at work on a 4-point scale ranging from 1 ("Strongly agree") to 4 ("Strongly disagree"). All items are summed. Potential scores range from 5-20, with higher scores indicative of lower levels of moral stress.
Adverse events | One week and 1, 3, and 6 month follow-up
  A free text response field measuring the occurrence of any health problems since the last contact.
Future self questionnaire - shortened version | 3 month follow-up
  A free text response field asking to imagine a future self identity. Then a free text response field to describe a mental image of this identity, 2 items measuring vividness (from 1 "not vivid at all" to 10 "very vivid") and positivity (from 1 "very negative" to 10 "very positive") of that image on a 10-point scale and 1 item measuring the perspective of viewing that mental image ("through own eyes" or "as if seeing oneself") before and after the traumatic event(s). Higher scores on rating scales indicate higher levels of vividness/positivity.
Time perspective questionnaire | Baseline (Day 1), One week, 1, 3, and 6 month follow-up
  8 self-report items (5-point scale from 1 to 5) measuring time perspective on three subscales: past perspective (items 3, 5, 7), present perspective (items 1, 8) and future perspective (items 2, 4, 6). Item scores for each subscale will be summed. Higher values indicate higher levels of past/present/future time perspective.
Coping mechanisms | Baseline (Day 1)
  2 free text response field questions (e.g. Are there any specific factors you think have made it easier for you to handle the COVID-19 situation and its consequences?) at Day 1.
WHODAS 2.0 | 6 month follow-up
  12 self-rated items assessing functioning in six life domains: 1) cognition, 2) mobility, 3) personal care 4) relations, 5) daily activities and 6) participation in society. Each item is rated on a 5-point scale, from 1 ("none") to 5 ("extreme or cannot do") and summed; a higher sum score indicates worse functioning. An additional three questions are asked at the end regarding the frequency and impact of these items.
Credibility/expectancy questionnaire | Day 1
  5 item questionnaire (11-point scale from 0 to 10) that rates to what degree the participant finds the intervention credible. High scores indicate greater credibility.
Subjective Units of Distress (SUDS) | Day 1
  A bespoke manipulation check item measuring self-rated distress during the intervention/control procedure (11-point scale from 0 to 10) at 3 times during the intervention process. Higher scores indicate higher level of distress.
Feedback questionnaire about participation | 1 month follow-up
  8 bespoke items including questions about study participation e.g. how acceptable was it to do the task? Rated on 11-point scale from 0 (not at all) to 10 (extremely), higher scores indicate higher acceptability; and questions about what has happened since the study with a yes/no response e.g. have you had any psychological or medical treatment since you did the task; and items with a free text response field e.g. do you have any other comments.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Holmes, Prof, Principal Investigator — Karolinska Institutet/Uppsala University
Locations (1):
- Hospital units across Sweden (e.g. FO Akut, Karolinska University Hospital Huddinge), Huddinge, Sweden

REFERENCES:
- [Derived] Kanstrup M, Singh L, Leehr EJ, Goransson KE, Pihlgren SA, Iyadurai L, Dahl O, Falk AC, Lindstrom V, Hadziosmanovic N, Gabrysch K, Moulds ML, Holmes EA. A guided single session intervention to reduce intrusive memories of work-related trauma: a randomised controlled trial with healthcare workers in the COVID-19 pandemic. BMC Med. 2024 Sep 19;22(1):403. doi: 10.1186/s12916-024-03569-8. PMID 39300443
- [Derived] Ahmed Pihlgren S, Johansson L, Holmes EA, Kanstrup M. Exploring healthcare workers' experiences of a simple intervention to reduce their intrusive memories of psychological trauma: an interpretative phenomenological analysis. Eur J Psychotraumatol. 2024;15(1):2328956. doi: 10.1080/20008066.2024.2328956. Epub 2024 Mar 27. PMID 38533843